CLINICAL TRIAL: NCT00784368
Title: A Pharmacokinetic Study of JK1211 in Patients With Systemic Fungal Infection (SFI) and Patients With Febrile Neutropenia (FN) Suspected of Fungal Infection.
Brief Title: A Pharmacokinetic Study of JK1211(Itraconazole [Itrizole]) Oral Solution in Participants With Deep Mycosis and Those With Febrile Neutropenia Suspected of Fungal Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR014299; JK1211-JPN-07 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2008-10-23; First posted 2008-11-03 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-06

CONDITIONS: Mycoses; Candidiasis; Aspergillosis; Cryptococcosis; Blastomycosis; Histoplasmosis; Neutropenia
Keywords: Mycoses; Candidiasis; Aspergillosis; Cryptococcosis; Blastomycosis; Histoplasmosis; Neutropenia; Itraconazole; JK1211
MeSH Terms: conditions — Mycoses; Candidiasis; Aspergillosis; Cryptococcosis; Blastomycosis; Histoplasmosis; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SFI (ITCZ Oral Solution Monotherapy) (Experimental): Participants with deep-seated mycosis (Systemic Fungal Infection [SFI]) received itraconazole (ITCZ) oral solution in the dose range of 20 milliliter (ml) per day to 40 ml per day for 12 weeks as per Investigator's discretion.
  Interventions: Drug: ITCZ Oral Solution
- SFI (Switched Treatment) (Experimental): Participants with SFI received 200 milligram (mg) twice daily itraconazole intravenous (into the vein) infusion (ITCZ-IV) for first 2 days followed by 200 mg per day ITCZ-IV up to 14 days. Participants then received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion.
  Interventions: Drug: ITCZ Oral Solution; Drug: ITCZ-IV
- FN (Switched treatment) (Experimental): Participants with febrile neutropenia (FN) with suspected fungal infection received 200 mg twice daily ITCZ-IV for first 2 days followed by 200 mg per day ITCZ-IV up to 14 days. Participants then received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion.
  Interventions: Drug: ITCZ Oral Solution; Drug: ITCZ-IV

INTERVENTIONS:
Drug: ITCZ Oral Solution — ITCZ syrup product containing ITCZ 10 mg per ml in dose range of 20 ml to 40 ml daily for 7 days up to 12 weeks
  Other Names: Itrizole Oral Solution 1%, JK1211
Drug: ITCZ-IV — 200 mg IV twice daily for 2 days and once daily for the next 1 to 12 days
  Arms: FN (Switched treatment); SFI (Switched Treatment)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) of itraconazole (ITCZ) oral solution in participants with Systemic Fungal Infection (SFI) and those with febrile (with fever) neutropenia (FN, decrease in white blood cells) suspected of fungal infection.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (conducted in more than 1 center) and uncontrolled (no competitive drugs involved) study. Participants with SFI will receive treatment with ITCZ oral solution or switch treatment from intravenous (into a vein) infusion of itraconazole (ITCZ-intravenous) to ITCZ oral solution as per Investigator's discretion. All the participants with FN suspected of fungal infection will receive the switch treatment from ITCZ- intravenous to ITCZ oral solution. The study will include 3 periods: Pre-observation period (7 days), Treatment period (85 days for ITCZ oral solution monotherapy and 99 days for switch treatment) and Follow-up observation period (30 days). The participants who receive ITCZ oral solution monotherapy will receive ITCZ oral solution without ITCZ-intravenous in the dose range of 20 milliliter (ml) per day to 40 ml per day for 12 weeks (85 days) and those on the switch treatment will receive 400 milligram (mg) per day ITCZ-intravenous twice for first 2 days followed by 200 mg per day ITCZ-intravenous up to 14 days and then they will be administered treatment as per ITCZ oral solution monotherapy. Efficacy will primarily be evaluated by assessing the pharmacokinetics. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* In case of participants with deep-seated mycosis (systemic fungal infection [SFI]) they should be either clinically suspected case or proven case
* All participants administered need to be hospitalized during the itraconazole intravenous treatment
* For participants with febrile (with fever) neutropenia (a decrease in white blood cells) suspected of fungal infection who have persistent fever (greater than equal to 37.5 degree celsius; greater than equal to 3 days) and have neutrophil count less than 500 per cubic millimeter (or less than 1000 per cubic millimeter and expected to decrease toward less than 500 per cubic millimeter

Exclusion Criteria:

* No past history of hypersensitivity to azole antifungal agents
* No current medication with antifungal agents such as amphotericin B (intravenous injection [injection of a substance into a vein], tablets, syrup), nystatin (tablets), fluconazole (capsules, intravenous injection), flucytosine (oral agent), miconazole (intravenous injection, gel), micafungin (intravenous infusion), fosfluconazole (intravenous injection,) voriconazole (intravenous injection, tablets), liposomal amphotericin B (intravenous injection), posaconazole
* No medication with itraconazole in any formulation within the last 28 days
* Participants with history of severe hepatic disease (except hepatic dysfunction because of fungal infection) and congestive heart failure
* Female participants who are either pregnant, nursing, suspected to be pregnant or will become pregnant during the trial duration

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K.,Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan

REFERENCES:
- See also: A Pharmacokinetics Study of JK1211 in Patient with "Deep Mycosis" and Those with "Febrile Neutropenia Suspected of Fungal Infection " — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=418&filename=CR014299_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- FN (Switched Treatment): Participants with febrile (with fever) neutropenia (a decrease in white blood cells) (FN) with suspected fungal infection received 200 mg twice daily ITCZ-IV for first 2 days followed by 200 mg per day ITCZ-IV up to 14 days. Participants then received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion.
Period: Overall Study
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment) | FN (Switched Treatment)
Started | 16 | 16 | 23
Completed | 8 | 5 | 12
Not Completed | 8 | 11 | 11
Not completed — Physician Decision | 0 | 0 | 6
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Adverse Event | 6 | 9 | 2
Not completed — Diagnosis of fever | 0 | 0 | 1
Not completed — Worsening of complications | 0 | 0 | 1
Not completed — Worsening of symptoms | 0 | 1 | 0
Not completed — Withdrawal of informed consent | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SFI (Switched Treatment): Participants with SFI received 200 milligram (mg) twice daily itraconazole intravenous infusion (ITCZ-IV) for first 2 days followed by 200 mg per day ITCZ-IV up to 14 days. Participants then received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment) | FN (Switched Treatment) | Total
Number analyzed (Participants) | 15 | 16 | 22 | 53
Age Continuous [Mean (Standard Deviation); unit: years] — Data for Baseline characteristic (Age) was available for 53 participants who were included in Full Analysis Set (FAS) population. FAS population included all participants except those who did not meet main eligibility criteria, who did not receive ITCZ-IV or ITCZ oral solution (ITCZ-OS) and participants without efficacy data. One participant without any infection evidence was not included in FAS for SFI (ITCZ OS Monotherapy).
  years | 61.7 (13.6) | 64.2 (12.0) | 58.3 (12.7) | 61.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Data for Baseline characteristic (Gender) was available for 53 participants who were included in FAS population. FAS population included all participants except those who did not meet main eligibility criteria, who did not receive ITCZ-IV or ITCZ-OS and participants without efficacy data. One participant without any infection evidence was not included in FAS for SFI (ITCZ OS Monotherapy).
  Participants
    Female | 1 | 6 | 7 | 14
    Male | 14 | 10 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Itraconazole Concentration (Cmax)
Description: The Cmax is defined as the maximum observed analyte concentration. Cmax was measured in microgram per milliliter (mcg/ml).
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: Pharmacokinetic (PK) analysis set included all participants who received ITCZ-OS and had plasma concentration data. One participant without any infection evidence was also included in the PK population for SFI (ITCZ-OS). 'n' signifies those participants who were evaluated for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 16 | 13 | 22
mcg/ml
  200 mg/day (n=11,5,12) | 2.90 (1.48) | 2.30 (1.12) | 1.79 (0.682)
  300 mg/day (n=4,2,0) | 9.20 (2.39) | 58.2 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported. | NA (NA) — No participant was administered 300 mg/day dose in the FN (Switched treatment) arm.
  400mg/day (n=1,6,10) | 0.948 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 6.10 (3.12) | 2.44 (0.996)

2. Primary Outcome: Area Under the Curve From Time Zero to 24 Hours Post-dose Observed Plasma Itraconazole Concentration (AUC[0-24])
Description: The AUC(0-24) is area under the plasma concentration time curve from time zero (pre-dose) to 24 hours post-dose. It is usually calculated by linear trapezoidal method. AUC was measured in mcg*hour(hr) per ml.
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: The PK analysis set included all participants who received ITCZ-OS and had plasma concentration data. One participant without any infection evidence was also included in the PK population, for SFI (ITCZ-OS). Here 'n' signifies those participants who were evaluated for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: mcg*hr per ml
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 16 | 13 | 22
mcg*hr per ml
  200 mg/day (n=11,5,12) | 55.8 (34.4) | 41.0 (25.6) | 31.4 (14.1)
  300 mg/day (n=4,2,0) | 207 (54.7) | 129 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported. | NA (NA) — No participant was administered 300 mg/day dose in the FN (Switched treatment) arm.
  400mg/day (n=1,6,10) | 19.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 137 (71.3) | 50.4 (23.5)

3. Primary Outcome: Minimum Inhibitory Concentration (MIC)
Description: The MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation.
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: The PK analysis set. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluated for this measure at specified time points for each arm group respectively. MIC was not obtained for FN (Switched treatment) and hence the data not given for the same.
Measure: Mean (Standard Deviation); unit: mcg per ml
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment)
Number analyzed (Participants) | 4 | 5
mcg per ml
  200 mg/day (n=4,1) | 0.438 (0.125) | 0.06 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  300 mg/day (n=0,1) | NA (NA) — No evaluable participant was treated with 300 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  400mg/day (n=0,3) | NA (NA) — No evaluable participant was treated with 400 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 0.71 (0.51)

4. Primary Outcome: Maximum Plasma Drug Concentration by Minimum Inhibitory Concentration (Cmax/MIC)
Description: The Cmax is maximum observed analyte concentration and MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. The Cmax/MIC was calculated only in participants for whom the MIC was obtained.
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment)
Number analyzed (Participants) | 4 | 5
ratio
  200 mg/day (n=4,1) | 7.21 (2.13) | 28.8 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  300 mg/day (n=0,1) | NA (NA) — No evaluable participant was treated with 300 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 5.81 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  400 mg/day (n=0,3) | NA (NA) — No evaluable participant was treated with 400 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 18.9 (21.6)

5. Primary Outcome: Area Under the Curve During 24 Hours by Minimum Inhibitory Concentration (AUC 0-24/MIC)
Description: The AUC (0-24) is defined as area under the plasma concentration-time curve over the dosing interval (24 hr). It is usually calculated by linear trapezoidal method. MIC is the lowest concentration of an antimicrobial that inhibits the visible growth of a microorganism after incubation. The AUC 0-24/MIC was calculated only in participants for whom the MIC was obtained.
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Groups:
- SFI (JK1211 Monotherapy): Participants with deep-seated mycosis (SFI) received JK1211 orally (taken by mouth; to be swallowed) in the dose range of 20 milliliter per day (ml/day) to 40 ml/day for 12 weeks as per Investigator's discretion.
Arm/Group | SFI (JK1211 Monotherapy) | SFI (Switched Treatment)
Number analyzed (Participants) | 4 | 5
hour
  200 mg/day (n=4,1) | 147 (56.6) | 399 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  300 mg/day (n=0,1) | NA (NA) — No evaluable participant was treated with 300 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 129 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  400 mg/day (n=0,3) | NA (NA) — No evaluable participant was treated with 400 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 421 (478)

6. Primary Outcome: Time Above Minimum Inhibitory Concentration (T>MIC)
Description: The T>MIC was calculated only in participants for whom the MIC was obtained.
Time Frame: Day 85 for SFI (ITCZ Oral Solution Monotherapy); and Day 99 for SFI and FN Switched treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment)
Number analyzed (Participants) | 4 | 5
percent time
  200 mg/day (n=4,1) | 100 (0) | 100 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  300 mg/day (n=0,1) | NA (NA) — No evaluable participant was treated with 300 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 100 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  400 mg/day (n=0,3) | NA (NA) — No evaluable participant was treated with 400 mg/day, so it was not possible to evaluate the relationship between the dose level and the pharmacokinetic parameters. | 100 (0)

7. Secondary Outcome: Number of Participants With Change in Clinical Symptoms by Centralized Assessment
Description: Level of improvement in the clinical symptoms was assessed as: disappeared (if clinical symptoms disappeared), improved (significant improvement in clinical symptoms ), no change (almost no improvement in the clinical symptoms), worsened (if the clinical symptoms worsened) and could not be assessed (if it was difficult to make the above-noted assessments).
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI and FN Switched treatment)
Population: FAS population included all participants except those who did not meet main eligibility criteria, who did not receive ITCZ-IV or ITCZ-OS and participants without efficacy data. As per planned analysis both SFI (ITCZ Oral Solution Monotherapy) and SFI (Switched Treatment) arms were combined for all efficacy analyses.
Measure: Number; unit: participants
Groups:
- SFI (ITCZ Oral Solution Monotherapy + Switched Treatment): Participants with SFI were allocated either to SFI (ITCZ Oral Solution Monotherapy) or SFI (Switched Treatment). Participants in SFI (ITCZ Oral Solution Monotherapy) group received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion. Participants in SFI (Switched Treatment) were administered 200 mg twice daily ITCZ-IV for first 2 days followed by 200 mg per day ITCZ-IV up to 14 days. Participants then received ITCZ oral solution in the dose range of 20 ml per day to 40 ml per day for 12 weeks as per Investigator's discretion.
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 31 | 22
participants
  Disappeared | 7 | 6
  Improved | 12 | 12
  No change | 7 | 2
  Worsened | 2 | 0
  Could not be assessed | 3 | 2

8. Secondary Outcome: Number of Participants With Change in Clinical Symptoms by Diagnosis Name (Centralized Assessment)
Description: Level of improvement in the clinical symptoms was assessed as: disappeared (if clinical symptoms disappeared), improved (significant improvement in clinical symptoms ), no change (almost no improvement in the clinical symptoms), worsened (if the clinical symptoms worsened) and could not be assessed (if it was difficult to make the above-noted assessments). The cases evaluated were candidemia, esophageal candidiasis, invasive aspergillosis, chronic necrotic pulmonary aspergillosis (C.N.P.A), pulmonary aspergilloma (P.A.) and pulmonary cryptococcosis (P.C).
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI Switched treatment)
Population: The FAS population. As per planned analysis both SFI arms were combined for efficacy analyses; participants with FN with suspected fungal infection were not planned to be analyzed for this outcome measure. Here, 'n' signifies those participants who were evaluated for this measure at specified time points for each arm group respectively.
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment)
Number analyzed (Participants) | 31
participants
  Candidemia: Improved (n=1) | 1
  Esophageal candidiasis: Disappeared (n=3) | 3
  Invasive aspergillosis: Disappeared (n=5) | 2
  Invasive aspergillosis: Improved (n=5) | 1
  Invasive aspergillosis: Worsened (n=5) | 1
  Invasive aspergillosis:Could not be assessed (n=5) | 1
  C.N.P.A: Improved (n= 8) | 5
  C.N.P.A: No change (n=8) | 3
  P.A.: Improved (n=10) | 4
  P.A.: No change (n=10) | 4
  P.A.: Could not be assessed (n=10) | 2
  P.C.: Disappeared (n=4) | 2
  P.C.: Improved (n=4) | 1
  P.C.: Worsened (n=4) | 1

9. Secondary Outcome: Percentage of Participants With Overall Response by Centralized Assessment
Description: Efficacy rate (E.R.) was calculated as number of cases for whom treatment was judged to be effective divided by sum of number of cases for whom treatment was judged to be effective and cases for whom treatment was judged to be ineffective multiplied by 100. Treatment success rate (T.S.R.) was calculated as number of cases for whom treatment was judged to be effective divided by sum of number of cases for whom treatment was judged to be effective, cases for whom treatment was judged to be ineffective and cases for whom the efficacy could not be assessed multiplied by 100.
Time Frame: as for outcome 7
Population: The FAS population included all participants except those who did not meet main eligibility criteria, who did not receive ITCZ-IV or ITCZ-OS and participants without efficacy data. As per planned analysis both SFI (ITCZ Oral Solution Monotherapy) and SFI (Switched Treatment) arms were combined for all efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 31 | 22
percentage of participants
  E.R. | 62.1 [42.3 to 79.3] | 80.0 [56.3 to 94.3]
  T.S.R | 58.1 [39.1 to 75.5] | 72.7 [49.8 to 89.3]

10. Secondary Outcome: Percentage of Participants With Overall Response by Diagnosis Name (Centralized Assessment)
Description: E.R. was calculated as number of cases for whom treatment was judged to be effective divided by sum of number of cases for whom treatment was judged to be effective and number of cases for whom treatment was judged to be ineffective multiplied by 100. T.S.R. was calculated as number of cases for whom treatment was judged to be effective divided by sum of number of cases for whom treatment was judged to be effective, number of cases for whom treatment was judged to be ineffective and number of cases for whom the efficacy could not be assessed multiplied by 100.
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI Switched treatment)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment)
Number analyzed (Participants) | 31
percentage of participants
  E.R.: Candidemia (n=1) | 100.0 [2.5 to 100]
  E.R.: Esophageal candidiasis (n=3) | 100.0 [29.2 to 100]
  E.R.: Invasive aspergillosis (n=5) | 60.0 [14.7 to 94.7]
  E.R.: C.N.P.A (n=8) | 62.5 [24.5 to 91.5]
  E.R.: P.A. (n=10) | 50.0 [15.7 to 84.3]
  E.R.: P.C. (n=4) | 50.0 [6.8 to 93.2]
  T.S.R. : Candidemia (n=1) | 100.0 [2.5 to 100]
  T.S.R. : Esophageal candidiasis (n=3) | 100.0 [29.2 to 100]
  T.S.R. : Invasive aspergillosis (n=5) | 60.0 [14.7 to 94.7]
  T.S.R. : C.N.P.A (n=8) | 62.5 [24.5 to 91.5]
  T.S.R. : P.A. (n=10) | 40.0 [12.2 to 73.8]
  T.S.R. : P.C. (n=4) | 50.0 [6.8 to 93.2]

11. Secondary Outcome: Number of Participants With Mycological Efficacy by Centralized Assessment
Description: Mycological efficacy was assessed as disappeared (if results for pathogenic fungus became negative, or if it was not possible to obtain the appropriate specimens), decreased (if level of pathogenic fungus was decreased in culture), no change (if there was no quantitative change in pathogenic fungus), increased (if there was a quantitative increase in pathogenic fungus, if results for pathogenic fungus became positive after start of dosing or if new pathogenic fungus was identified) , could not be assessed (if it was difficult to make the above assessment due to lack of detection in tests).
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 31 | 22
participants
  Disappeared | 6 | 0
  No change | 1 | 0
  Could not be assessed | 24 | 22

12. Secondary Outcome: Number of Participants With Mycological Efficacy by Diagnosis Name (Centralized Assessment)
Description: Mycological efficacy was assessed as disappeared, decreased, no change, increased, could not be assessed. The cases evaluated were candidemia, esophageal candidiasis, invasive aspergillosis, C.N.P.A, P.A. and P.C.
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI Switched treatment)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment)
Number analyzed (Participants) | 31
participants
  Candidemia: Could not be assessed (n=1) | 1
  Esophageal candidiasis: Disappeared (n=3) | 1
  Esophageal candidiasis:Could not be assessed (n=3) | 2
  Invasive aspergillosis:Could not be assessed (n=5) | 5
  C.N.P.A: Disappeared (n=8) | 1
  C.N.P.A: No change (n=8) | 1
  C.N.P.A: Could not be assessed (n=8) | 6
  P.A.: Disappeared (n=10) | 3
  P.A.: Could not be assessed (n=10) | 7
  P.C.: Disappeared (n=4) | 1
  P.C.: Could not be assessed (n=4) | 3

13. Secondary Outcome: Number of Participants With Serological Effect Against Fungi by Centralized Assessment
Description: Serological effect against fungi was assessed as changed to negative (if the test values became negative), improved (if the test values decreased), no change (if there was no change in the test values), no change (if there was no change in the test values) , worsened (if the test values increased) and could not be assessed (if it was difficult to make the above-noted assessments due to a reason such as a lack of detection in the tests before and after dosing).
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 31 | 22
participants
  Changed to negative | 1 | 0
  Improved | 3 | 0
  No change | 5 | 1
  Worsened | 2 | 2
  Could not be assessed | 20 | 19

14. Secondary Outcome: Number of Participants With Serologic Effect Against Fungi by Diagnosis Name (Centralized Assessment)
Description: Serological effect against fungi was assessed as changed to negative (if the test values became negative), improved (if the test values decreased), no change (if there was no change in the test values), worsened (if the test values increased) and could not be assessed (if it was difficult to make above-noted assessments due to a reason such as a lack of detection in the tests before and after dosing). The cases evaluated were candidemia, esophageal candidiasis, invasive aspergillosis, C.N.P.A, P.A. and P.C.
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI Switched treatment)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment)
Number analyzed (Participants) | 31
participants
  Candidemia: Changed to negative (n=1) | 1
  Esophageal candidiasis:Could not be assessed (n=3) | 3
  Invasive aspergillosis: No change (n=5) | 1
  Invasive aspergillosis: Worsened (n=5) | 1
  Invasive aspergillosis:Could not be assessed (n=5) | 3
  C.N.P.A: Improved (n=8) | 2
  C.N.P.A: Worsened (n=8) | 1
  C.N.P.A: Could not be assessed (n=8) | 5
  P.A.:No change (n=10) | 1
  P.A.: Could not be assessed (n=10) | 9
  P.C.: Improved (n=4) | 1
  P.C.: No change (n=4) | 3

15. Secondary Outcome: Number of Participants With Change In the Endoscopy or Image Diagnosis By Centralized Assessment
Description: Level of Improvement in the Endoscopy or Image diagnosis was assessed as disappeared (if the abnormal findings were normalized), decreased (if level of pathogenic fungus was decreased in culture), improved (if significant improvement was observed in the abnormal findings), no change (if no significant improvement was observed in the abnormal findings), worsened (if the abnormal findings were worsened) and could not be assessed (if it was difficult to make the above-noted assessments due to a reason such as a lack of detection in the tests before and after dosing).
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment) | FN (Switched Treatment)
Number analyzed (Participants) | 31 | 22
participants
  Disappeared | 3 | 0
  Improved | 12 | 0
  No change | 7 | 0
  Worsened | 4 | 1
  Could not be assessed | 5 | 21

16. Secondary Outcome: Number of Participants With Change in the Endoscopy or Image Diagnosis by Diagnosis Name (Centralized Assessment)
Description: Level of Improvement in Endoscopy was assessed as disappeared, decreased, improved, no change, worsened and could not be assessed. The cases evaluated were candidemia, esophageal candidiasis, invasive aspergillosis, C.N.P.A, P.A. and P.C.
Time Frame: Baseline up to end of treatment (Day 85 for SFI [ITCZ Oral Solution Monotherapy] and Day 99 for SFI Switched treatment)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | SFI (ITCZ Oral Solution Monotherapy + Switched Treatment)
Number analyzed (Participants) | 31
participants
  Candidemia: Could not be assessed (n=1) | 1
  Esophageal candidiasis: Disappeared (n=3) | 3
  Invasive aspergillosis: Improved (n=5) | 3
  Invasive aspergillosis: Worsened (n=5) | 2
  C.N.P.A: Improved (n=8) | 3
  C.N.P.A: No change (n=8) | 3
  C.N.P.A: Worsened (n=8) | 2
  P.A.:Improved (n=10) | 3
  P.A.:No change (n=10) | 4
  P.A.: Could not be assessed (n=10) | 3
  P.C.: Improved (n=4) | 3
  P.C.: Could not be assessed (n=4) | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug
Arm/Group | SFI (ITCZ Oral Solution Monotherapy) | SFI (Switched Treatment) | FN (Switched Treatment)
Serious Adverse Events (participants affected / at risk) | 4/16 | 8/16 | 3/23
Other Adverse Events (participants affected / at risk) | 15/16 | 16/16 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SFI (ITCZ Oral Solution Monotherapy) (N=16) | SFI (Switched Treatment) (N=16) | FN (Switched Treatment) (N=23)
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aplastic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tremors (Nervous system disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Kidney damage (Renal and urinary disorders) | 1 | 0 | 0
Edema (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SFI (ITCZ Oral Solution Monotherapy) (N=16) | SFI (Switched Treatment) (N=16) | FN (Switched Treatment) (N=23)
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6 | 12
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 8
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 10 | 6
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 5 | 4 | 10
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Renal disorder (Renal and urinary disorders) | 3 | 2 | 2
Renal tubular disorder (Renal and urinary disorders) | 2 | 2 | 2
Oedema (General disorders) | 0 | 3 | 3
Oedema peripheral (General disorders) | 2 | 2 | 1
Beta 2 microglobulin urine increased (Investigations) | 7 | 7 | 5
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 4 | 2 | 5
Alpha 1 microglobulin urine increased (Investigations) | 3 | 3 | 2
Blood cholesterol decreased (Investigations) | 1 | 2 | 4
C-reactive protein increased (Investigations) | 4 | 1 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 5
Platelet count decreased (Investigations) | 2 | 2 | 2
Urine analysis abnormal (Investigations) | 2 | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 0
Blood glucose increased (Investigations) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.